CLINICAL TRIAL: NCT03873220
Title: Feasibility for Quantification of Scratch Behavior and Sleep in Children With Atopic Dermatitis
Brief Title: Monitoring Of Scratch Via Accelerometry In Children
Acronym: MOSAIC
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: H-37801
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Atopic Dermatitis
Keywords: Wearable devices; Scratch; Sleep
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monitoring scratch in children: Sensor technology and digital measures will be used to evaluate scratch and sleep in children with atopic dermatitis who will wear watch-like wrist actigraphy devices, sleep monitor, polysomnography, and videography.
  Interventions: Device: Wrist Actigraphy Devices; Device: Sleep Monitor; Device: Polysomnography; Device: Videography

INTERVENTIONS:
Device: Wrist Actigraphy Devices — A watch-like wearable sensor
  Other Names: GENEActiv Watch
Device: Sleep Monitor — Remote Sensor
  Other Names: EarlySense
Device: Polysomnography — Sleep Monitor
Device: Videography — Thermal Camera

SUMMARY:
Sleep sensors, wrist worn accelerometers, polysomnography (PSG), and associated data analysis platforms would provide quantitative and qualitative knowledge regarding the action of scratching and sleep quantity in a symptomatic atopic dermatitis (AD) population. The overall aim of this research is to validate the use of sensor technology and digital measures to quantitatively and qualitatively evaluate scratch and sleep in AD patients, and specifically in this study in children ages 2 to 11 years. To evaluate this experimental paradigm, the investigators propose using wearable accelerometers, a sleep sensor, PSG, videography and associated traditional patient-reported outcome measures/clinical outcome assessments (PRO/COA) in patients/caregivers with AD in a well-controlled in-laboratory and at-home study.

DETAILED DESCRIPTION:
To assess the feasibility of quantifying scratch and sleep in children with Atopic Dermatitis (AD), children, age 2 to 11 years, with AD will be recruited. The subjects will complete specific questionnaires related to itch, sleeping habits and AD and continuously wear two wrist worn accelerometry devices. The EarlySense Sleep Monitor will also be placed underneath the mattress to measure additional sleep related activities.

The study will be comprised of two overnight sleep laboratory site visits. The clinic visits will be followed by a continuous ~48 hour in-home environment assessment period (defined as the subject's daily routine environment). During the sleep lab site visit, the subject and accompanying parent(s)/guardian(s) will sleep overnight at the facility. The subject will be video-recorded during the in-sleep lab visit, wear the wrist accelerometry devices, use the sleep sensor and complete assessments (Depending on age, parent/guardian may complete some assessments). Upon the completion of sleep lab activities the subjects will then continue to wear the wrist accelerometry devices, utilize the sleep sensor and complete Patient Reported Outcome/Clinical Outcome Assessments (PRO/COA) assessments during the 48 hour in-home assessment. At the conclusion of the in-home portion of the assessment, the subject will return the device/s and assessments to the facility and undergo brief assessments/interview.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥2 years of age and <12 years of age at Day 1.
2. Written informed consent from parent(s)/guardian(s) and assent from the subject (where assent is applicable).
3. Native English speakers or demonstrated fluency in English (both subject and parent(s)/guardian(s)).
4. Has a clinical diagnosis of Atopic Dermatitis (AD) according to the criteria of Hanifin and Rajka (concomitant AD treatments are permitted on study).

Exclusion Criteria:

1. AD affected surface areas are in a location of device placement.
2. Has unstable AD (Total BSA>40%).
3. Has any planned surgical or medical procedure that would overlap with study participation.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Individuals diagnosed with atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Quantification of scratch using GENEActiv watches to assess triaxial accelerometry | From enrollment through the end of visit 5 (5 days +/- 2 days).
  One GENEActiv watch will be used on each hand at a sampling rate of 100 Hz to measure movement in the x, y, and z direction. The movement will be analyzed using the algorithm described by Cole et al. to differentiate between periods of wakefulness and sleep.
Quantification of sleep using Polysomnography | From enrollment through the end of visit 5 (5 days +/- 2 days).
  Polysomnography (PSG) will be used to report the number of sleep occurrences and appropriate sleep staging based on the scoring guide provided by the American Academy of Sleep Medicine (AASM) for children. The following sleep stages will be scored: Stage W (wakefulness), Stage N1 (NREM 1), Stage N2 (NREM 2), Stage N3 (NREM 3), Stage N (NREM), and Stage R (REM).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD MBA, Principal Investigator — Boston University, Department of Anatomy and Neurobiology
Locations (1):
- Evans Biomedical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided